CLINICAL TRIAL: NCT05573100
Title: A Randomized, Open-label, Parallel-group, Multi-center Phase 2a Study to Evaluate the Efficacy and Safety of CU06-1004 for 12 Weeks in Patients With Diabetic Macular Edema (DME)
Brief Title: The Study of CU06-1004 in Patients With Diabetic Macular Edema (DME)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Curacle Co., Ltd. (Industry)
Collaborators: Théa Open Innovation, France (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CU06-RE-P2A-01
Record Dates: First submitted 2022-09-25; First posted 2022-10-10 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2023-07

CONDITIONS: Diabetic Macular Edema
Keywords: DME; Endothelial dysfunction blocker
MeSH Terms: interventions — CU06-1004

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CU06-1004 100mg (Experimental): CU06-1004 100 mg tablets. Dosed at 100 mg (1 capsule) QD within 30 minutes after meal on each evening
  Interventions: Drug: CU06-1004
- CU06-1004 200mg (Experimental): CU06-1004 100 mg tablets. Dosed at 200 mg (2 capsules) QD within 30 minutes after meal on each evening
  Interventions: Drug: CU06-1004
- CU06-1004 300mg (Experimental): CU06-1004 100 mg tablets. Dosed at 300 mg (3 capsules) QD within 30 minutes after meal on each evening
  Interventions: Drug: CU06-1004

INTERVENTIONS:
Drug: CU06-1004 — CU06-1004 per capsule for oral administration. CU06-1004 is a white off powder at room temperature. The CU06-1004 100 mg soft gelatin capsules consist of a solution-based fill.
  Other Names: SAC-1004; CU06; CU06-RE

SUMMARY:
This phase 2a trial is a randomized, open-label, parallel-group study in approximately 60 patients with DME to evaluate the efficacy and safety of CU06-1004 orally administered once daily for 12 weeks. The study will have a 1:1:1 randomization (CU06-1004 100mg: CU06-1004 200mg: CU06-1004 300mg).

ELIGIBILITY:
Inclusion Criteria:

1. Subject who is male or female ≥ 18 years of age
2. Subject who has a diagnosis of Type 1 or 2 diabetes mellitus
3. Subject who has study eye with definite retinal thickening due to diabetic macular edema involving the center of the macula
4. Subject who has voluntarily signed an informed consent form
5. Subject who has study eye with central subfield thickness (CST) of the following on SD-optical coherence tomography (OCT).

   1. Zeiss Cirrus: CST ≥ 290 µm in women, or ≥ 305 µm in men
   2. Heidelberg Spectralis: CST ≥ 305 µm in women, or ≥ 320 µm in men
6. Subject who has DRSS score ≥ 35
7. Subject who has study eye with an ETDRS BCVA letter score ranging from 34 to 83, inclusive (approximate Snellen equivalent of 20/25 - 20/200 at a distance of 4 meters).
8. Subject who has media clarity, pupillary dilation, and subject cooperation sufficient for adequate fundus photographs.

Exclusion Criteria:

1. Subject whose macular edema is of non-diabetic retinopathy etiology (e.g., secondary to vitreomacular interface abnormalities).
2. Subject who has had major surgery within 3 months prior to randomization or major surgery planned during the next 6 months.
3. Subject who has a hypersensitivity to any excipients of the investigational product or similar class of drug and ingredient.
4. Subject who has the following illness or abnormal laboratory test values:

   * Uncontrolled hypertension (SBP > 180 mmHg or DBP > 100 mmHg)
   * Uncontrolled diabetes (HbA1c > 12.0%)
   * Total bilirubin > 1.5 × ULN
   * Positive results for HIV or Hepatitis B or C viruses
   * Other clinically significant abnormal lab values per Investigator's judgement
5. Subject who participated in an investigational trial of biologic agent within 3 months and any other investigational trial within 1 month of randomization.
6. Subject who has received gene therapy for any indication.
7. Subject who has received COVID-19 vaccine within 30 days of first dosing until the end of the study.
8. Pregnant woman, lactating woman, or female or male subject of childbearing potential who doesn't accept appropriate contraceptive measures for the next 6 months

   * Hormonal contraceptives, intrauterine contraceptive device, sterilization of spouse (e.g., vasectomy, tubal ligation), double-barrier method (e.g., combinational use of spermicides and condoms, diaphragm, contraceptive sponge, or FemCap)
9. Subject who has medical condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure, cardiovascular disease, and glycemic control).
10. Subject who administered vaccinium myrtillus extract or dobesilate calcium within 2 weeks before randomization.
11. Subject who has unstable angina, myocardial infarction, transient ischemic attack, cerebral infarction, coronary artery bypass surgery, or transluminal coronary angioplasty within 6 months before screening.
12. Subject who has an ocular condition (other than diabetes) that, in the opinion of the investigator, might affect macular edema or alter visual acuity during the course of the study (e.g., vein occlusion, uveitis or other ocular inflammatory disease, neovascular glaucoma, Irvine-Gass Syndrome, foveal atrophy, pigmentary changes, dense subfoveal hard exudates, nonretinal condition etc.).
13. Subject who has exam evidence of external ocular infection, including conjunctivitis, chalazion, or significant blepharitis.
14. Subject who is expected to have no improvement of decreased visual acuity in the opinion of the Investigator, even if macular edema is resolved (e.g., foveal atrophy, abnormal pigmentation, dense subfoveal hard exudate).
15. Subject who has a history of treatment with anti-VEGF agents, or focal laser treatment (Focal/grid laser photocoagulation) within 3 months prior to randomization or intravitreal dexamethasone or triamcinolone within 6 months prior to randomization.
16. Subject who has a history of treatment with intravitreal fluocinolone astonide.
17. Subject who has a history of panretinal scatter photocoagulation (PRP).
18. Subject who anticipated need for PRP in the 3 months following randomization.
19. Subject who has a history of ocular surgery (including cataract extraction, any intraocular surgery, etc.) within prior 3 months or anticipated within the next 6 months following randomization.
20. Subject who has a history of retinal detachment or retinal detachment repair surgery.
21. Subject who has a history of YAG capsulotomy performed within 2 months prior to randomization.
22. Subject who has uncontrolled glaucoma in either eye (intraocular pressure (IOP) > 24 mmHg on medication or according to the investigator's judgment).
23. Subject who has a history of vitrectomy.
24. Subject who has any active intraocular inflammatory diseases such as uveitis, conjunctivitis, and in either eye.
25. Subject who has any history of intraocular inflammation in either eye other than what would be expected in the normal post-operative course following prior routine ocular surgery such as cataract surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2022-12-21 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
The change of central subfield thickness (CST) | Baseline and 12 weeks
  Change in CST in the study eye assessed by SD-OCT at Week 12 compared to baseline
To determine the optimal doses | 12 weeks
  The 1:1:1 randomization is fitting for the study objective to determine the optimal doses for a phase 2b study.

SECONDARY OUTCOMES:
The change of central subfield thickness (CST) | Baseline, 4 weeks and 8 weeks
  Change in CST in the study eye assessed by SD-OCT Weeks 4 and 8 compared to baseline
The change of all other subfield thickness | Baseline, 4 weeks, 8 weeks and 12 weeks
  Change in all other subfield thickness (Nasal, temporal, superior and inferior) in the study eye assessed by SD-OCT at Weeks 4, 8, and 12 compared to baseline
The change of early treatment diabetic retinopathy study (ETDRS) best-corrected visual acuity (BCVA) letter score | Baseline, 4 weeks, 8 weeks and 12 weeks
  Change in ETDRS BCVA letter score in the study eye at Weeks 4, 8, and 12 compared to baseline
Change in diabetic retinopathy severity scale (DRSS) | Baseline and 12 weeks
  Change in DRSS in the study eye at Weeks 12 compared to baseline
The change of blood biomarkers | Baseline and 12 weeks
  Change in blood biomarker (TNF-alpha, IL-1 beta, IL-6) at Week 12 compared to baseline
Number and severity of treatment emergent adverse events (TEAEs) | Baseline and 12 weeks
  Number and severity of TEAEs up to Week 12 compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Pankyung Kim, M.S, Study Director — Curacle Co., Ltd.
Locations (11):
- United States (10):
  - Rand Eye Institute, Deerfield Beach, Florida
  - Elman Retina Group, Baltimore, Maryland
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - New England Retina Consultants, Springfield, Massachusetts
  - Mid Atlantic Retina, Bethlehem, Pennsylvania
  - Austin Research Center for Retina, Austin, Texas
  - Retina consultant of Texas, Bellaire, Texas
  - Valley Retina Institute, McAllen, Texas
  - Wagner Macula and Retina Center, Norfolk, Virginia
- Emanuelli Research & Development Center, Arecibo, Puerto Rico

IPD SHARING:
Plan to Share IPD: No